CLINICAL TRIAL: NCT05405075
Title: Arizona Alzheimer's Disease Research Center (ADRC)
Status: Recruiting | Type: Observational
Sponsor: Banner Health (Other)
Responsible Party: Sponsor
Other Study IDs: ADRC-001
Record Dates: First submitted 2022-03-04; First posted 2022-06-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Arizona Alzheimer's Disease Research Center (ADRC) is the National Institute on Aging's (NIA's) first statewide AD Center (ADC), the only ADC in the Southwestern United States, and a leading example of statewide collaboration in biomedical research. It capitalizes on Arizona's strengths in brain imaging, genomics, computer science and biomathematics, the basic, cognitive and behavioral neurosciences, clinical, and neuropathological studies of AD, the discovery and evaluation of investigational treatments, and the study of normal cognitive aging.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal persons, individuals with mild cognitive impairment or dementia who are at least 40 years of age.
* Willing to undergo health and cognitive assessments, and collection and banking of blood with venipuncture for genetic research, biomarker research, and DNA banking.

Exclusion Criteria:

* 1. Participants whose diagnosis is unclear and confounded by multiple possible factors are excluded. Participants with diagnoses of non-AD dementias are not excluded.

  2. Participants whose primary diagnosis is cognitive impairment due to a penetrating or single severe closed head injury, multiple sclerosis, brain tumor, metabolic or toxic encephalopathy, post-infectious (e.g., viral encephalitis, bacterial meningitis), paraneoplastic, primary psychiatric illness, or otherwise not deemed relevant to the intent of the Alzheimer Disease Center program are excluded.

  3. Procedure specific exclusion criteria also apply but this does not impact the participants ability to be included in the study.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Clinical Core maintains a target of 550 participants at all stages of the aging-dementia spectrum including 400 normal controls and 150 participants with MCI, probable AD dementia and other dementias. Embedded within these diagnostic categories are defined Latino and Native American cohorts.
  Participants will be referred to the ADRC from varying sources including, but not limited to, clinic referrals, community outreach programs, general advertising, national registries, and other sites within the consortium.
  Participants eligible for enrollment and those completing annual follow-up are discussed in frequent diagnostic consensus conferences. All undergo a standardized neuropsychological and neurological battery of tests at entry and annual tests at all sites.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Status | 12 months
  The ADRC uses a prospective, standardized, and longitudinal clinical evaluation of participants to determine their cognitive status. This includes tests that assess short and long term memory, ability to complete daily tasks, and processing of information.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Banner Alzheimer's Institute - Tucson, Tucson, Arizona